CLINICAL TRIAL: NCT04069728
Title: The Impact of 3D Anal Fistula Models on Patient Understanding and Decision Making
Acronym: 3DAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RD19/027
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2020-12

CONDITIONS: Fistula in Ano; Ano Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: Prospective randomised pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard clinic appointment (Other): Patients who undergo a routine clinic outpatient appointment using standard explanation of their fistula with words, diagrams and MRI images, as per Consultant preference
  Interventions: Other: Standard explanation
- Clinic appointment with 3D model (Experimental): Patients who undergo a routine clinic outpatient appointment using a 3D printed model to assist explanation of their fistula
  Interventions: Other: Explanation with 3D printed fistula model

INTERVENTIONS:
Other: Explanation with 3D printed fistula model — Explanation of fistula and surgery using a 3D printed model of an anal fistula that depicts the anatomy of the anal canal, the path of the anal fistula and its relation to anatomic structures.
  Arms: Clinic appointment with 3D model
Other: Standard explanation — Explanation of fistula and treatment using words, diagrams and MRI images as per consultant choice. Standard clinical care.
  Arms: Standard clinic appointment

SUMMARY:
An anal fistula is an abnormal communication between the luminal surface of the anorectal canal and the perianal skin. Fistulas can vary in their complexity and can be challenging to treat, due to the anatomical relation to the anal sphincter complex that controls continence. In addition, fistulas can display complex features such as branches, cavities and horseshoes; where the tract travels radially around the anal canal. All these features have a role in determining the most appropriate surgical treatment option, and are key to understanding the surgical decision-making process. This study will determine patient understanding of fistula anatomy, their perception of their own understanding, their rating of how good their clinician's explanation is and how this impacts the decision-making process using standard explanation with 2D images, versus a 3D printed model of a fistula.

DETAILED DESCRIPTION:
Previous work has established a method of using traditional two-dimensional MR images to construct and print 3D models of perianal fistula, however the clinical utility of these models in the outpatient setting and their impact on patient knowledge of disease have not yet been assessed. This study is aimed at understanding how the use of 3D printed models can influence patient understanding of disease and support them in making decisions regarding treatment.

Participants attending routine outpatient appointments will have their fistula explained to them using either a standard explanation, or a 3D printed model of a fistula. They will complete a short series of questionnaires and their answers will be analysed to determine if there is any benefit of using 3D models in a clinical consultation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Aged ≥18 years old
* Patients who are new referrals to complex fistula clinic
* Patients with an idiopathic or Crohn's perianal fistula
* Patients with an intersphincteric or transsphincteric fistula according to Park's classification
* Patients who have had MR imaging of their anal fistula prior to consultation
* Able to give full informed consent

Exclusion Criteria:

Patients < 18 years

* Patients with a rectovaginal or pouch fistula
* Fistula secondary to malignancy or radiation
* Suprasphincteric or extrasphincteric fistulas
* Follow up patients
* Patients who have no prior MR imaging of their fistula Patients who do not have the capacity to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Patient understanding of fistula anatomy and surgery | 5 minutes
  A score obtained using a non-validated questionnaire that assesses the patient's understanding of their fistula anatomy and the treatment that has been proposed.
  Scores can range from 0 to 16, with a higher score suggesting better understanding.

SECONDARY OUTCOMES:
Patient understanding of their fistula: Patient reported subjective assessment | 1 minute
  A self reported score that patients give for how well they feel they have understood their fistula and proposed surgery. Patients rate how well they understand their fistula on a scale of 1-10, where 1 denotes very poor understanding, and 10 equates to excellent understanding.
Quality of explanation: Patient reported subjective assessment | 1 minute
  Patient reported subjective rating of how well their clinician explained their fistula and surgery to them. Four questions where patients rate how well their fistula was explained on a scale of 1 to 10, with 1 equating to very poor understanding and 10 excellent understanding. An additional question asks the patient if the explanation relieved their anxiety (Yes/No). Responses to individual questions will be reported.
Decisional Conflict Scale | 5 minutes
  A validated questionnaire that assesses the level of uncertainty a patient has in making a decision. Subscales:
  Uncertainty: Scores range from 0 (feels extremely certain) to 100 (feels extremely uncertain about best choice) Informed: Scores range from 0 (feels extremely informed) to 100 (extremely uninformed) Values clarity: Scores range from 0 (feels clear about personal values for benefits and risks) to 100 (feels extremely unclear about personal values) Support: Scores range from 0 (feels extremely supported in decision making) to 100 (feels unsupported in decision making) Effective decision: Scores range from 0 (good decision) to 100 (bad decision). The total score is obtained by the addition of each individual score, which is then divided by 16 and multiplied by 25. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict)
3D model utility | 1 minute
  Patient reported subjective rating of how useful the 3D model was, using a non- validated questionnaire. This includes 3 questions where patients rate how useful the model is on a scale of 1 to 10, with 1 equating to not very useful, and 10 being very useful. The final question asks patients if they would like to see models in future consultations (Yes/No). Responses to individual questions will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Mr Tozer, Principal Investigator — LONDON NORTH WEST UNIVERSITY HEALTHCARE NHS TRUST
Locations (1):
- London North West University Healthcare NHS Trust, Harrow, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biglino G, Koniordou D, Gasparini M, Capelli C, Leaver LK, Khambadkone S, Schievano S, Taylor AM, Wray J. Piloting the Use of Patient-Specific Cardiac Models as a Novel Tool to Facilitate Communication During Cinical Consultations. Pediatr Cardiol. 2017 Apr;38(4):813-818. doi: 10.1007/s00246-017-1586-9. Epub 2017 Feb 18. PMID 28214968
- [Background] Sahnan K, Adegbola SO, Tozer PJ, Patel U, Ilangovan R, Warusavitarne J, Faiz OD, Hart AL, Phillips RKS, Lung PFC. Innovation in the imaging perianal fistula: a step towards personalised medicine. Therap Adv Gastroenterol. 2018 May 24;11:1756284818775060. doi: 10.1177/1756284818775060. eCollection 2018. PMID 29854001
- [Background] Bernhard JC, Isotani S, Matsugasumi T, Duddalwar V, Hung AJ, Suer E, Baco E, Satkunasivam R, Djaladat H, Metcalfe C, Hu B, Wong K, Park D, Nguyen M, Hwang D, Bazargani ST, de Castro Abreu AL, Aron M, Ukimura O, Gill IS. Personalized 3D printed model of kidney and tumor anatomy: a useful tool for patient education. World J Urol. 2016 Mar;34(3):337-45. doi: 10.1007/s00345-015-1632-2. Epub 2015 Jul 11. PMID 26162845
- [Background] Roy M, Novak CB, Urbach DR, McCabe SJ, von Schroeder HP, Okrainec K. Decisional conflict in surgical patients: Should surgeons care? Can J Surg. 2019 Mar 22;62(3):1-3. Online ahead of print. PMID 30900439
- [Background] Sander IM, Liepert TT, Doney EL, Leevy WM, Liepert DR. Patient Education for Endoscopic Sinus Surgery: Preliminary Experience Using 3D-Printed Clinical Imaging Data. J Funct Biomater. 2017 Apr 7;8(2):13. doi: 10.3390/jfb8020013. PMID 28387702
- [Derived] Iqbal N, Fletcher J, Bassett P, Hart A, Lung P, Tozer P. Exploring methods of improving patient understanding and communication in a complex anal fistula clinic: results from a randomized controlled feasibility study. Colorectal Dis. 2024 Mar;26(3):518-526. doi: 10.1111/codi.16861. Epub 2024 Jan 18. PMID 38235831
- See also: Decisional conflict scale questionnaire and user manual — https://decisionaid.ohri.ca/eval_dcs.html